CLINICAL TRIAL: NCT05740969
Title: Gene and Protein Expression Profiles After Treatment of Actinic Keratoses
Acronym: PACKS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ismail Gögenur (Other)
Responsible Party: Sponsor-Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG-163-2021
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; Imiquimod; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5-Fluorouracil (Active Comparator): Patients will be asked apply a 40 mg/g creme containing 5-Fluorouracil once a day on their lesion for 10 days. A biopsy will be taken four days after last application. The patient will be refered to a dermatologist for further treatment, if necessary.
  Interventions: Drug: 5Fluorouracil
- Imiquimod (Active Comparator): Patients will be asked apply a 50 mg/g creme containing imiquimod thrice a week on their lesion for 10 days. A biopsy will be taken four days after last application. The patient will be refered to a dermatologist for further treatment, if necessary.
  Interventions: Drug: Imiquimod
- Melatonin (Experimental): Patients will be asked apply a 25 mg/g creme containing melatonin once a day on their lesion for 10 days. A biopsy will be taken four days after last application. The patient will be refered to a dermatologist for further treatment, if necessary.
  Interventions: Drug: Melatonin
- Control (No Intervention): A biopsy will be taken from the patient and the patient will be refered to a dermatologist for further treatment, if necessary.

INTERVENTIONS:
Drug: 5Fluorouracil — Cream
  Arms: 5-Fluorouracil
Drug: Imiquimod — Cream
  Arms: Imiquimod
Drug: Melatonin — Cream
  Arms: Melatonin

SUMMARY:
The primary aim of this study is to investigate the effect of 5-fluorouracil, imiquimod, and melatonin for actinic keratosis on immunological gene, and protein expressions profiles. Secondarily, the aim is to assess the effect of the treatment on the histopathology of actinic keratoses.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have a clinical diagnosis of actinic keratosis
* Participants should be 18 years old or above
* Participants must sign an informed consent

Exclusion Criteria:

* Known allergic reaction to either 5-fluorouracil , imiquimod, or melatonin
* Immunomodulating treatment
* Predictable poor compliance (due to i.e. dementia, substance abuse, psychiatric disease, life-threatening disease or language barriers)
* Pregnant or breastfeeding
* Females not in menopause (defined as no menstruation during the last 12 months) should use a secure birth control (intrauterine devices, hormonal contraceptives including - oral pills, patches, vaginal rings and injections) during the entire period of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gene and protein expression profiles | 10 days of treatment

SECONDARY OUTCOMES:
histopathological assessment of actinic keratoses | 10 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ismail A. Gögenur, MD, DMSc, Principal Investigator — Center For Surgical Science, Dept. of Surgery, Zealand University Hosptial
Locations (1):
- Zealand University Hospital, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No